CLINICAL TRIAL: NCT02559804
Title: Prospective Study Registry of Peripheral Neuroblastic Tumours Presenting With Spinal Canal Involvement (SCI)
Acronym: NB-SCI
Status: Recruiting | Type: Observational
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Collaborators: Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor
Other Study IDs: NB with SCI
Record Dates: First submitted 2015-09-11; First posted 2015-09-24 (Estimated); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Neuroblastic Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients NB with SCI: Survival and late effects. Diagnosis of peripheral neuroblastic tumour - peripheral neuroblastic tumour (neuroblastoma, ganglioneuroblastoma, ganglioneuroma) presenting with SCI, symptomatic or asymptomatic, independent of disease extension (stage), and clinical course (first diagnosis or relapse/progression).
  Interventions: Other: survival and late effects

INTERVENTIONS:
Other: survival and late effects — survival and late effects

SUMMARY:
To describe the natural history of peripheral neuroblastic tumour presenting with SCI and evaluate the combined effects of different risk factors on the eventual neurologic and orthopaedic outcomes

DETAILED DESCRIPTION:
Multi-centre, observational, prospective study registry. About 15% of patients with peripheral neuroblastic tumour present with extradural SCI, of whom approximately 60% are symptomatic. Since SCI may progress to irreversible paraplegia, early diagnosis and prompt treatment is of critical importance.1-3 The treatment options include chemotherapy, neurosurgical decompression and radiation therapy. All may relieve epidural compression, but there is no consensus on which to use first in the individual patient. However, the choice of the treatment could be relevant in the perspective of reducing to the minimum the risk of long-term sequelae.4 Guidelines for the diagnostic work-up and treatment of SCI for International Society of Paediatric Oncology European Neuroblastoma (SIOPEN) neuroblastoma patients were already available in the "guidelines for the treatment of patients with localized resectable neuroblastoma and analysis of prognostic factors" (LNESG1 Protocol), back in 1994,5 although it is unknown how they were applied in the SIOPEN Centres. These guidelines have been reformulated in occasion of the recently activated "European Low and Intermediate risk Neuroblastoma" (LINES Protocol).

There are few publications addressing the diagnosis and treatment of SCI; most are retrospective studies, case reports, or reviews that may be affected by reporting bias.1-9 Therefore new guidelines could be designed based on the information derived from a prospective data collection of newly diagnosed patients.

For this study Spinal Canal Involvement (SCI) is defined when, referring to an axial plane of the spinal cord MRI scan (Figure 1), the tumour extends into the vertebral canal and goes beyond a mentally drown ellipsoid (red circle) passing through the cortical bone of both anterior and posterior arches of the vertebra. This involvement is called "intraspinal" or, better, "intracanal".

Patient data to be collected and included in the corresponding Forms

1. work-up at diagnosis, including radiology report (Computed Tomography or Magnetic Resonance Imaging)
2. treatment administered
3. response to treatment, including radiology report
4. follow-up
5. outcome

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of peripheral neuroblastic tumour - peripheral neuroblastic tumour (neuroblastoma, ganglioneuroblastoma, ganglioneuroma) presenting with SCI, symptomatic or asymptomatic, independent of disease extension (stage), and clinical course (first diagnosis or relapse/progression)
* No previous chemotherapy, except steroids, in the last 6 months
* Age <18 years
* Minimal planned follow-up of 5 years
* Parent/patient written informed consent (Appendix 1(A,B,C))

Exclusion Criteria:

* Invasion of intervertebral foramina only

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients in the age range 0-18 years diagnosed with peripheral neuroblastic tumour and SCI in the period from May 2014 to April 2017
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-05; Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of neurologic consequences | for 5 years
  American Spinal Injury Association ASIA impairment scale
prevalence of orthopedic consequences | for 5 years
  using Common Terminology Criteria for Adverse Events v. 4.0
prevalence of pain | for 5 years
  using Face, Legs, Activity, Cry, Consolability scale (FLACC scale)

SECONDARY OUTCOMES:
relapse or second tumour | 5 years
  event free survival
survival | 5 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Haupt, MD, Principal Investigator — Istituto Giannina Gaslini Genova
Locations (1):
- Istituto Giannina Gaslini, Genova, Italy